CLINICAL TRIAL: NCT05311059
Title: Impact of Laparoscopic Ovarian Drilling on Ovarian Reserve (Serum Anti-mullerian Hormone Levels - Antral Follicular Count and Ovarian Volume) in Patients With Anovulatory Polycystic Ovarian Syndrome
Brief Title: Impact of Laparoscopic Ovarian Drilling on Ovarian Reserve in Patients With Anovulatory Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64
Record Dates: First submitted 2022-03-08; First posted 2022-04-05 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian drilling (Experimental): Drilling needle was introduced and connected by monopolar current, held against ovarian surface for 4 seconds using a power of 40 watt, 4 puncture was done in each ovary with putting into consideration that the puncture must be not superficial and it must go deep through the main substance of the ovary
  Interventions: Procedure: Laparoscopic ovarian drilling

INTERVENTIONS:
Procedure: Laparoscopic ovarian drilling — Drilling needle was introduced and connected by monopolar current, held against ovarian surface for 4 seconds using a power of 40 watt, 4 puncture was done in each ovary with putting into consideration that the puncture must be not superficial and it must go deep through the main substance of the ovary

SUMMARY:
Pneumoperitoneum is done by insertion of the verress needle at the inferior edge of the umbilicus putting into consideration the following tests:

1. Needle test: Verress needle patency check.
2. Hissing phenomenon: Needle introduced by open valve mechanism.
3. Aspiration test: Placing a drop of water on the opening of the needle and examine its disappearance into the abdomen.
4. Volume test: Changes occurred in the intra abdominal pressure during gas insufflations.

Intra abdominal pressure 12-16 mmHg usually suitable for this pelvic surgery. Introduction of the laparoscopic instruments all in its place

* Laparoscopic telescope : From the inferior edge of umbilicus through trocar and sleeve which inserted by corkscrew technique then removed to allow the telescope insertion which connected to light source , camera head and color monitor.
* 2nd and 3rd punctures were done allowing another two graspers to be inserted usually at a point represent outer 1/3 of the lateral abdominal wall in an imaginary line from umbilicus to iliac bone

Puncturing technique :

Fixation of one ovary away from intestine by grasping the ovarian ligament with the traumatic grasper which allow good exposure of the ovary and allow drilling .

Drilling needle was introduced and connected by monopolar current, held against ovarian surface for 4 seconds using a power of 40 watt, 4 puncture was done in each ovary with putting into consideration that the puncture must be not superficial and it must go deep through the main substance of the ovary.

Cooling of the ovary by lactated ringer's solution, finally removal of all instruments under vision after exclusion of any complication .

DETAILED DESCRIPTION:
Pneumoperitoneum is done by insertion of the verress needle at the inferior edge of the umbilicus putting into consideration the following tests:

1. Needle test: Verress needle patency check.
2. Hissing phenomenon: Needle introduced by open valve mechanism.
3. Aspiration test: Placing a drop of water on the opening of the needle and examine its disappearance into the abdomen.
4. Volume test: Changes occurred in the intra abdominal pressure during gas insufflations.

Intra abdominal pressure 12-16 mmHg usually suitable for this pelvic surgery. Introduction of the laparoscopic instruments all in its place

* Laparoscopic telescope : From the inferior edge of umbilicus through trocar and sleeve which inserted by corkscrew technique then removed to allow the telescope insertion which connected to light source , camera head and color monitor.
* 2nd and 3rd punctures were done allowing another two graspers to be inserted usually at a point represent outer 1/3 of the lateral abdominal wall in an imaginary line from umbilicus to iliac bone.

Puncturing technique :

Fixation of one ovary away from intestine by grasping the ovarian ligament with the traumatic grasper which allow good exposure of the ovary and allow drilling .

Drilling needle was introduced and connected by monopolar current, held against ovarian surface for 4 seconds using a power of 40 watt, 4 puncture was done in each ovary with putting into consideration that the puncture must be not superficial and it must go deep through the main substance of the ovary.

Cooling of the ovary by lactated ringer's solution, finally removal of all instruments under vision after exclusion of any complication .

ELIGIBILITY:
Inclusion Criteria:

* o Age of woman: 18 - 35 y.

  * Anovulatory PCO.
  * Clomiphene citrate resistant Woman:
* Full dose of Clomiphene citrate.
* 6 Months of ovarian induction.

  * Normal semen analysis and Hystrosalpingography

Exclusion Criteria:

* o Age below 18y or above 35.

  * Ovulatory PCO.
  * Responder to Clomiphene citrate.
  * Obvious cause of infertility rather than PCO.
  * Hyperandrogenism due to any other endocrinal disorder

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
Antral follicular count | 3 months from laparoscopy
  AFC is defined as counting of all echo lucent rounded follicles measuring (2-10mm) that present in the substance of the ovary
AntiMullerian hormone | 3 months from laparoscopy
  Plasma samples were assayed for AMH in duplicate using a commercial enzyme-linked immunosorbant assay kit.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided